CLINICAL TRIAL: NCT04514653
Title: A Phase 2, Randomized, Dose-escalation, Ranibizumab-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of RGX-314 Gene Therapy Delivered Via One or Two Suprachoroidal Space (SCS) Injections in Participants With Neovascular Age-Related Macular Degeneration (nAMD) (AAVIATE)
Brief Title: RGX-314 Gene Therapy Administered in the Suprachoroidal Space for Participants With Neovascular Age-Related Macular Degeneration (nAMD)
Acronym: AAVIATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RGX-314-2102 (M23-411); M23-411 (Other: AbbVie Inc)
Record Dates: First submitted 2020-08-04; First posted 2020-08-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD)
Keywords: AMD; wet AMD; wAMD; nAMD
MeSH Terms: interventions — Ranibizumab; Piperacillin, Tazobactam Drug Combination; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The vision examiners and central reading center (CRC) graders will be masked, meaning they will be unaware of the participants' treatment assignment. All other individuals affiliated with the study (investigators, all study center personnel apart from the vision examiners, the participants, all staff of Sponsor and its research collaborator, all staff affiliated with the contract research organization, and all CRC staff apart from the CRC graders) will have knowledge of the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (7):
- Ranibizumab control (Active Comparator): Control treatment arm
  Interventions: Biological: Ranibizumab
- ABBV-RGX-314 Treatment Arm (Dose 1) (Experimental): ABBV-RGX-314 Dose 1
  Interventions: Genetic: ABBV-RGX-314 Dose 1
- ABBV-RGX-314 Treatment Arm (Dose 2) (Experimental): ABBV-RGX-314 Dose 2
  Interventions: Genetic: ABBV-RGX-314 Dose 2
- ABBV-RGX-314 Treatment Arm (Dose 3) (Experimental): ABBV-RGX-314 Dose 3
  Interventions: Genetic: ABBV-RGX-314 Dose 3
- ABBV-RGX-314 Treatment Arm (Dose 3) and Local Steroid (Experimental): ABBV-RGX-314 Dose 3 and Local Steroid
  Interventions: Genetic: ABBV-RGX-314 Dose 3; Drug: Local Steroid
- ABBV-RGX-314 Treatment Arm (Dose 3) and Topical Steroid (Experimental): ABBV-RGX-314 Dose 3 and Topical Steroid
  Interventions: Genetic: ABBV-RGX-314 Dose 3; Drug: Topical Steroid
- ABBV-RGX-314 Treatment Arm (Dose 4) and Topical Steroid (Experimental): ABBV-RGX-314 Dose 4 and Topical Steroid
  Interventions: Drug: Topical Steroid; Genetic: ABBV-RGX-314 Dose 4

INTERVENTIONS:
Biological: Ranibizumab — Ranibizumab (anti-VEGF agent)
  Arms: Ranibizumab control
Genetic: ABBV-RGX-314 Dose 1 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 1)
  Other Names: Combination Product
  Arms: ABBV-RGX-314 Treatment Arm (Dose 1)
Genetic: ABBV-RGX-314 Dose 2 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 2)
  Other Names: Combination Product
  Arms: ABBV-RGX-314 Treatment Arm (Dose 2)
Genetic: ABBV-RGX-314 Dose 3 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 3)
  Other Names: Combination Product
  Arms: ABBV-RGX-314 Treatment Arm (Dose 3); ABBV-RGX-314 Treatment Arm (Dose 3) and Local Steroid; ABBV-RGX-314 Treatment Arm (Dose 3) and Topical Steroid
Drug: Local Steroid — Local steroid
  Arms: ABBV-RGX-314 Treatment Arm (Dose 3) and Local Steroid
Drug: Topical Steroid — Topical steroid
  Arms: ABBV-RGX-314 Treatment Arm (Dose 3) and Topical Steroid; ABBV-RGX-314 Treatment Arm (Dose 4) and Topical Steroid
Genetic: ABBV-RGX-314 Dose 4 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 4)
  Other Names: Combination Product
  Arms: ABBV-RGX-314 Treatment Arm (Dose 4) and Topical Steroid

SUMMARY:
This interventional study is being conducted with an investigational gene therapy treatment called ABBV-RGX-314 (also known as RGX-314) and is being developed as a potential one-time gene therapy treatment for neovascular (wet) age-related macular degeneration (wet AMD or nAMD). The typical treatment for nAMD is frequent injections of anti-VEGF therapy. Researchers are testing ABBV-RGX-314 to see if it has similar effects as the current approved standard of care, such as Lucentis® or Eylea® injections.

The duration of this study will be up to 52 weeks or for ranibizumab control participants who cross over to ABBV-RGX-314 after week 52, up to 80 weeks post-randomization.

The primary outcome measure for this investigational study is to evaluate the mean change in best-corrected visual acuity (BCVA) for ABBV-RGX-314 compared with ranibizumab monthly at the Week 40 visit.

DETAILED DESCRIPTION:
This phase 2, randomized, dose-escalation study is designed to evaluate the efficacy, safety and tolerability of ABBV-RGX-314 gene therapy in subjects with nAMD.

ABBV-RGX-314 will be injected into the SCS part of the eye. Approximately 140 participants who meet the inclusion/exclusion criteria will be enrolled into one of 7 cohorts. Participants will be randomized in Cohorts 1 and 2 to receive ABBV-RGX-314 or the intravitreal ranibizumab control. Participants enrolled in Cohorts 3 through 5 will receive ABBV-RGX-314. Participants enrolled in Cohort 6 will receive ABBV-RGX-314 and will be randomized to one of two different post-procedural steroid regimens. Participants randomized in Cohort 7 will receive ABBV-RGX-314 with a protocol mandated steroid regimen or the intravitreal ranibizumab control. Cohort 1 will evaluate ABBV-RGX-314 Dose 1, Cohorts 2 and 3 will evaluate ABBV-RGX-314 Dose 2, Cohorts 4, 5, and 6 will evaluate ABBV-RGX-314 Dose 3, and Cohort 7 will evaluate ABBV-RGX-314 Dose 4.

The duration of the study will be up to 52 weeks or for ranibizumab control participants who cross over to ABBV-RGX-314, up to 80 weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 50 and </= 89
* Diagnosis of CNV secondary to age-related macular degeneration in the study eye.
* Participants must have demonstrated a meaningful response to anti-VEGF therapy.
* Willing and able to provide written, signed informed consent for this study.

Exclusion Criteria:

* CNV or macular edema in the study eye secondary to any causes other than AMD.
* Subfoveal fibrosis or atrophy in study eye.
* Participants who have had a prior vitrectomy.
* Active or history of retinal detachment in the study eye.
* History of intravitreal therapy in the study eye, such as intravitreal steroid injection or investigational product (IP), other than anti-VEGF therapy, in the 6 months prior to study entry.
* Received any gene therapy.
* Any condition preventing visualization of the fundus or VA improvement in the study eye, eg, cataract.
* History of intraocular surgery in the study eye within 12 weeks of study entry.
* Receipt of any IP within 30 days of study entry or 5 half-lives of the IP.
* Myocardial infarction, cerebrovascular accident, or transient ischemic attacks within 6 months of study entry.
* Cohorts 1 - 5 only: Uncontrolled glaucoma in the study eye.

COHORT 6 AND 7 ONLY:

* Active or history of glaucoma or ocular hypertension (steroid-induced ocular hypertension (Cohort 7 only)) in the study eye.
* Certain OCT characteristics including: Large Pigment Epithelial Detachments (PED), clinically significant Epiretinal Membrane (ERM) in the study eye at Visit 1.

Note: Other inclusion/exclusion criteria apply.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA to Week 40 based on the Early Treatment Diabetic Retinopathy Study (ETDRS) score | 40 weeks
  The scale used is the early treatment diabetic retinopathy study (ETDRS) letter score from 0-100 and higher score being better vision.

SECONDARY OUTCOMES:
Incidence of overall and ocular adverse events (AEs) and serious adverse events (SAEs) | 52 weeks
  Incidence of overall and ocular adverse events (AEs) and serious adverse events (SAEs)
Vector shedding analysis in serum, urine, and tears | 52 Weeks
  Evaluate the safety and tolerability of ABBV-RGX-314
Proportion of participants who experience ocular inflammation following SCS ABBV-RGX-314 administration | 52 weeks
  To evaluate the incidences of ocular inflammation following SCS ABBV-RGX-314 administration
Mean change from baseline in choroidal neovascularization (CNV) lesion size and leakage area based on fluorescein angiography (FA) | Up to Week 80
  To evaluate the effect of ABBV-RGX-314 on CNV lesion growth and leakage as measured by FA
Mean change from baseline in BCVA based on ETDRS score | Up to Week 80
  Evaluate the effect of ABBV-RGX-314 on BCVA
Proportion of participants (1) gaining ≥ 15, ≥ 10, ≥ 5, or ≥ 0 letters; (2) losing ≥ 15, ≥ 10, ≥ 5, or > 0 letters (3) maintaining vision (not losing ≥ 15 letters) compared with baseline as per BCVA | Up to Week 52
  To evaluate the effect of ABBV-RGX-314 on BCVA
Mean change from baseline in CRT as measured by SD-OCT | Up to Week 80
  To evaluate the effect of ABBV-RGX-314 on CRT, as measured by SD-OCT
Mean supplemental anti-VEGF injection annualized rate in the ABBV-RGX-314 treatment arms | Up to Week 80
  To assess the need for supplemental anti-VEGF therapy in participants who receive ABBV-RGX-314 treatment
Proportion of participants who have a reduction of ≥ 50% and ≥ 75% in supplemental anti-VEGF- injection annualized rate | 52 Weeks
  Proportion of participants who have a reduction of ≥ 50% and ≥ 75% in supplemental anti-VEGF- injection annualized rate through Week 40 and Week 52 compared with the prior 52 weeks preceding the first intravitreal ranibizumab injection received as part of the Screening Period (ABBV-RGX-314 administered participants)
Proportion of participants with 0, ≤ 1, and ≤ 2 supplemental injections | Up to Week 80
  To assess the need for supplemental anti-VEGF therapy in participants who receive ABBV-RGX-314 treatment
Mean percent reduction in supplemental anti-VEGF injection annualized rate | Up to Week 80
  To assess the need for supplemental anti-VEGF therapy in participants who receive ABBV-RGX-314 treatment
Time from ABBV-RGX-314 administration to first supplemental anti-VEGF injection | 80 Weeks
  To assess the need for supplemental anti-VEGF therapy in participants who receive ABBV-RGX-314 treatment
Aqueous humor ABBV-RGX- 314 TP concentration over time | 52 Weeks
  To evaluate the concentration of ABBV-RGX-314 TP in aqueous humor and serum
Mean change from baseline in serum ABBV-RGX-314 TP concentration over time | 80 Weeks
  To evaluate the concentration of ABBV-RGX-314 TP in aqueous humor and serum

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- United States (18):
  - Retinal Research Institute /ID# 255925, Phoenix, Arizona
  - California Retina Consultants - Bakersfield /ID# 255910, Bakersfield, California
  - Retina Vitreous Assoc Med Grp /ID# 255921, Beverly Hills, California
  - Retinal Diagnostic Center /ID# 272275, Campbell, California
  - Northern California Retina Vitreous Associates Medical Group, Inc /ID# 255920, Mountain View, California
  - Retina Consultants of San Diego /ID# 255911, Poway, California
  - California Retina Consultants - Santa Barbara /ID# 255923, Santa Barbara, California
  - Southeast Retina Center /ID# 255912, Augusta, Georgia
  - Springfield Clinic - First /ID# 272274, Springfield, Illinois
  - Johns Hopkins Hospital /ID# 255919, Baltimore, Maryland
  - Ophthalmic Consultants of Boston /ID# 255917, Boston, Massachusetts
  - Sierra Eye Associates /ID# 255908, Reno, Nevada
  - Eye Associates of New Mexico /ID# 255915, Albuquerque, New Mexico
  - Duke University Medical Center /ID# 267646, Durham, North Carolina
  - Mid Atlantic Retina /ID# 255906, Philadelphia, Pennsylvania
  - Charles Retina Institute /ID# 255922, Germantown, Tennessee
  - Tennessee Retina - Nashville /ID# 255918, Nashville, Tennessee
  - Retina Consultants - The Woodlands /ID# 255924, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=RGX-314-2102